CLINICAL TRIAL: NCT02183974
Title: Suitable Method for Routine Diagnostics of EER in Children With Otitis Media With Effusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FNO-ENT-OME Restech
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Otitis Media With Effusion
Keywords: otitis media with effusion; Laryngopharyngeal Reflux
MeSH Terms: conditions — Otitis Media with Effusion; Laryngopharyngeal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peptest (Experimental): 44 children at the age between 1 to 7 years diagnosed with bilateral or unilateral OME who underwent adenoidectomy and myringotomy with insertion of ventilation tube. Effusion was collected and analysed using Peptest, which contains monoclonal antibodies targeted against pepsin. Result of the Peptest was stated as positive (2 lines), negative (1 line) and invalid (no line).
  Interventions: Procedure: Peptest

INTERVENTIONS:
Procedure: Peptest

SUMMARY:
The aim of the study was detection of pepsin in effusion in children with OME using Peptest as new quick and cheap method of detection and comparison results with results of other studies in which pepsin was detected by more demanding methods. Such a type of study hasn't been done so far.

DETAILED DESCRIPTION:
Children at the age between 1 to 7 years diagnosed with bilateral or unilateral OME who underwent adenoidectomy and myringotomy with insertion of ventilation tube were included in the prospective study. OME was defined as effusion in the middle ear behind intact eardrum longer than 3 months. Diagnosis was made on the basis of otomicroscopic findings, pneumatic otoscopy, type B tympanometry and audiometry (in older cooperative children). Children with no fluid in middle ear during myringotomy were revised as having tympanosclerosis and were excluded from the study. Children with craniofacial abnormities (Down syndrome, Treacher Collins syndrome, clefts etc.) were excluded from the study, as well. Demographic data and symptoms of EER disease were provided by parents, who were particularly inquired regarding the hoarseness, recurrent lower respiratory infection (bronchitis, pneumonia) and bronchial asthma of their child.

Myringotomy using microscope was done in anterior inferior part of the tympanic membrane. Type of middle ear effusion (fluid, mucous) was registered. Middle ear fluid was collected by special suction device with collecting bottle and ventilation tube was inserted in the tympanic membrane. In case of bilateral OME, effusion was collected and analysed separately. Specimen was first standardized. An amount of 0.1 ml of 10 % citric acid was added, specimen was centrifuged for 10 minutes and subsequently original migration reagent was added. Afterwards, specimen was examined using Peptest, which contains monoclonal antibodies targeted against pepsin. Result of the Peptest was stated as positive (2 lines), negative (1 line) and invalid (no line). Peptest detection limit is 16ng/ml of pepsin. Statistical analysis was done using MS Excel.

ELIGIBILITY:
Inclusion Criteria:

* signing of the informed consent
* children at the age between 1 to 7 years diagnosed with bilateral or unilateral OME

Exclusion Criteria:

* children with craniofacial abnormities (Down syndrome, Treacher Collins syndrome, clefts etc.)

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2012-06; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The frequency of the presence of pepsin in effusion in the middle ear as an indirect diagnostic method of extraesophageal reflux in children with otitis media with effusion | 2 years
  The frequency of the presence of pepsin in effusion in the middle ear was detected using Peptest in children with OME

CONTACTS AND LOCATIONS:
Overall Officials: Martin Formánek, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

REFERENCES:
- [Background] Zelenik K, Matousek P, Urban O, Schwarz P, Starek I, Kominek P. Globus pharyngeus and extraesophageal reflux: simultaneous pH <4.0 and pH <5.0 analysis. Laryngoscope. 2010 Nov;120(11):2160-4. doi: 10.1002/lary.21147. PMID 20938965
- [Background] He Z, O'Reilly RC, Mehta D. Gastric pepsin in middle ear fluid of children with otitis media: clinical implications. Curr Allergy Asthma Rep. 2008 Nov;8(6):513-8. doi: 10.1007/s11882-008-0094-7. PMID 18940143
- [Background] O'Reilly RC, He Z, Bloedon E, Papsin B, Lundy L, Bolling L, Soundar S, Cook S, Reilly JS, Schmidt R, Deutsch ES, Barth P, Mehta DI. The role of extraesophageal reflux in otitis media in infants and children. Laryngoscope. 2008 Jul;118(7 Part 2 Suppl 116):1-9. doi: 10.1097/MLG.0b013e31817924a3. PMID 18594333